CLINICAL TRIAL: NCT02341456
Title: A Phase Ib, Dose Finding Study Evaluating AZD1775 in Monotherapy, in Combination With Carboplatin and Paclitaxel, and in Combination With Only Carboplatin in Adult Asian Patients With Advanced Solid Tumours
Brief Title: Phase Ib Study AZD1775 in Combination With Carboplatin and Paclitaxel in Adult Asian Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6011C00003
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Advanced Solid Tumours
MeSH Terms: interventions — adavosertib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD1775 (Experimental): AZD1775 will be administered orally as a single dose on Day 1 Cycle 0. Following a 5±2 days washout period, AZD1775 (5 doses BID over 2.5 days) will be taken in combination with paclitaxel and carboplatin in each 21-day cycle for 6 cycles. Following 6 cycles of combination treatment, patients may continue on AZD1775 monotherapy (5 doses BID Day 1 to Day 2.5 in each 21-day cycle) at the investigator's discretion.
  Interventions: Drug: AZD1775
- Paclitaxel (Experimental): Commercially available paclitaxel will be administered at a dosage of 175 mg/m2 as a 3-hour IV infusion on Cycle Day 1 of a 21-day cycle for 6 cycles.
  Interventions: Drug: Paclitaxel
- Carboplatin (Experimental): Following the paclitaxel infusion, carboplatin will be administered at a dose of AUC 5 as an IV infusion on Cycle Day 1 of a 21-day cycle for 6 cycles. According to the Cancer Therapy Evaluation Program Information Letter Regarding the AUC Based Dosing of Carboplatin, the maximum carboplatin dose should not exceed the target AUC (mg*min/mL)*150 mL/min, but it may be less (Ivy et al 2010). For this study, the maximum dose of carboplatin cannot exceed a total dose of 750 mg.
  Interventions: Drug: carboplatin

INTERVENTIONS:
Drug: AZD1775 — AZD1775 is a highly selective, adenosine-triphosphate (ATP) competitive, small-molecule inhibitor of the WEE1 kinase that sensitizes tumour cells to cytotoxic agents and is being developed for the treatment of advanced solid tumours and p53 pathway deficient malignancies. Gemcitabine is a nucleoside analog used as chemotherapy.
  Other Names: MK1775
  Arms: AZD1775
Drug: Paclitaxel — Paclitaxel is a mitotic inhibitor used in cancer chemotherapy ; it and docetaxel represent the taxane family of drugs.
  Arms: Paclitaxel
Drug: carboplatin — Carboplatin is a chemotherapy drug used against some forms of cancer (mainly ovarian carcinoma, lung, head and neck cancers as well as endometrial, esophageal, bladder, breast and cervical; central nervous system or germ cell tumors; osteogenic sarcoma, and as preparation for a stem cell or bone marrow transplant.).
  Arms: Carboplatin

SUMMARY:
This is a phase Ib, open-label, multicentre study of AZD1775 administered orally in monotherapy and in combination with carboplatin and paclitaxel to Asian patients with advanced solid tumours.

DETAILED DESCRIPTION:
This is a phase Ib, open label, multicentre study of AZD1775 administered orally in monotherapy and in combination with carboplatin and paclitaxel in Asian patients with advanced solid tumours. The study design allows escalation or de-escalation of AZD1775 in combination with carboplatin and paclitaxel with intensive safety monitoring to ensure the safety of the patients. Approximately 12 evaluable patients will be enrolled in the dose-finding portion of this study. The total number of patients will depend upon the number of combination dose level evaluations necessary to define the recommended dose for further clinical evaluation. The proposed combination doses are : Dose level-1; Dose level 1; Dose level 2 (if Dose Level 1 tolerated). All combination doses other than Combination Dose level 1 may be subject to change by the SRC in light of emerging data. At least 3 and up to 6 evaluable patients will be required for each dose finding cohort. Once the recommended dose for further clinical evaluation is established, additional 3 to 6 patients may be enrolled to the cohort where the recommended dose has been defined to further characterise the safety, tolerability, pharmacokinetics, and efficacy profiles of AZD1775 in combination with paclitaxel and carboplatin. If this dose is subsequently found to be non-tolerated, alternative doses and/or schedules may be explored. This will be determined by the SRC.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of a locally advanced or metastatic solid tumour, excluding lymphoma, that failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
* At least 1 measureable lesion that can be accurately assessed at baseline by computerised tomography (CT) or magnetic resonance imaging (MRI) for solid tumours assessed using RECIST v1.1.
* World Health Organisation performance status 0 to 1 with no deterioration over the previous 2 weeks and a minimum life expectancy of ≥12 weeks.

Exclusion Criteria:

* Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days (if investigational agent does not have well characterised PK profile) or 5 × half-lives of the first dose of study treatment
* Patient has had prescription or non-prescription drugs or other products (ie, grapefruit juice) known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors or inducers of CYP3A4, which cannot be discontinued 2 weeks before Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug. Co-administration of aprepitant during this study is prohibited.
* AZD1775 is an inhibitor of breast cancer resistance protein (BCRP). The use of statins including Atorvastatin which are substrates for BCRP are therefore prohibited and patients should be moved on to non-BCRP alternatives.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Paul De Souza, MD, Principal Investigator — Liverpool Hospital, New South Wales; Dr. Jason Lickliter, MD, Principal Investigator — Nucleus Network Limited, Victoria; Dr. Noboru Yamamoto, MD, Principal Investigator — NCC Hospital; Dr Toshihiko Doi, MD, Principal Investigator — NCC Hospital (East); Prof Yung Ju Bang, Principal Investigator — Seoul National University Hospital; Prof Sang Prof Sang, Principal Investigator — Asan Medical Centre; Prof Keunchil Park, Principal Investigator — Samsung Medical Centre
Locations (5):
- Australia (2):
  - Research Site, Liverpool
  - Research Site, Melbourne
- Japan (2):
  - Research Site, Kashiwa
  - Research Site, Sapporo
- Research Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 clinical investigational sites located in Australia (2), Japan (2), and South Korea (3). A total of 21 subjects consented and 19 were enrolled between January 14, 2015 and June 13, 2016.
Pre-assignment Details: Total 21 subjects were consented to participate in the study. One (1) subject was screen failure, and one (1) other subject withdrew prior to treatment; Nineteen (19) subjects received treatment under the protocol.
Groups:
- Cohort 1: Subjects in Cohort 1 received a single oral dose of 175 mg of AZD1775 monotherapy followed 5 ± 2 days later by combination therapy consisting of 5 oral doses of 175 mg AZD1775 given 12 hours apart on days 1, 2, and 3 and single doses of intravenous paclitaxel (175 mg/m²) and intravenous carboplatin (AUC 5) given on day 1 of 21 day cycles.
- Cohort 1a: Subjects in Cohort 1a received a single oral dose of 175 mg of AZD1775 monotherapy followed 5 ± 2 days later by combination therapy consisting of 5 oral doses of 175 mg AZD1775 given 12 hours apart on days 1, 2, and 3 and single doses of intravenous carboplatin (AUC 5) given on day 1 of 21 day cycles.
- Cohort 2: Subjects in Cohort 2 received a single oral dose of 225 mg of AZD1775 monotherapy followed 5 ± 2 days later by combination therapy consisting of 5 oral doses of 225 mg AZD1775 given 12 hours apart on days 1, 2, and 3 and single doses of intravenous paclitaxel (175 mg/m²) and intravenous carboplatin (AUC 5) given on day 1 of 21 day cycles.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Started | 7 | 6 | 6
Completed | 3 | 0 | 2
Not Completed | 4 | 6 | 4
Not completed — Disease progression | 2 | 3 | 1
Not completed — Death | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Moved to local access programme. | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population is comprised of all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2 | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 5 | 18
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (5.23) | 43.0 (14.10) | 52.2 (13.82) | 50.3 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 11
  Male | 4 | 3 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 6 | 6 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Australia | 2 | 0 | 0 | 2
  Japan | 3 | 1 | 1 | 7
  Korea, Republic Of | 2 | 5 | 5 | 12
Smoking History [Count of Participants; unit: Participants]
  Never Used Tobacco | 4 | 4 | 3 | 11
  Former Smoker | 3 | 2 | 2 | 7
  Current Smoker | 0 | 0 | 1 | 1
Cancer Diagnosis [Count of Participants; unit: Participants]
  Head and Neck | 2 | 0 | 0 | 2
  Other; Gallbladder | 1 | 0 | 0 | 1
  Stomach | 1 | 0 | 0 | 1
  Cervix | 1 | 1 | 0 | 2
  Ovary | 1 | 0 | 1 | 2
  Uterus | 1 | 0 | 1 | 2
  Breast | 0 | 1 | 3 | 4
  Pancreas | 0 | 1 | 0 | 1
  Other; Thymic | 0 | 2 | 0 | 2
  Skin/Soft Tissue | 0 | 1 | 0 | 1
  Lung | 0 | 0 | 1 | 1
Type of Tobacco Product Used [Count of Participants; unit: Participants]
  Cigarettes | 3 | 2 | 3 | 8
  Cigars | 0 | 0 | 0 | 0
  Cigarillo | 0 | 0 | 0 | 0
  No history of tobacco use | 4 | 4 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events
Description: The number of patients with treatment-emergent adverse events was analyzed on the safety analysis set which was comprised of all patients who received at least one dose of the investigational drug.
Time Frame: Up to 21 days (1 Cycle)
Population: All patients who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 6 | 6
Participants
  Patients with ≥ 1 Adverse Event (AE) | 7 | 6 | 6
  Patients with ≥ 1 Treatment-Emergent AE (TEAE) | 6 | 6 | 6
  Patients with TEAE Related to Treatment | 6 | 4 | 6
  Patients with Serious TEAE | 3 | 0 | 4
  Patients with Severe TEAE | 6 | 4 | 6
  Patients with TEAE with AZD1775 discontinued | 1 | 0 | 2
  Patients with TEAE with paclitaxel discontinued | 1 | NA — Patients in Cohort 1a did not receive paclitaxel. | 2
  Patients with TEAE with carboplatin discontinued | 0 | 0 | 2
  Patients with TEAE and fatal outcome | 1 | 0 | 1
  Patients with Dose-Limiting Toxicity | 1 | 1 | 2

2. Primary Outcome: Number of Treatment-Emergent Adverse Events (TEAE)
Description: The number of treatment-emergent adverse events was counted in the safety analysis set which was comprised of all patients who received at least one dose of the investigational drug.
Time Frame: Up to 21 days (1 Cycle)
Population: All patients who received at least one dose of the investigational drug.
Measure: Number; unit: TEAE
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 6 | 6
TEAE
  Number of Adverse Events (AEs) | 370 | 202 | 382
  Number of TEAEs | 362 | 182 | 381
  Number of TEAEs Related to Study Treatment | 262 | 95 | 263
  Number of Serious TEAEs | 9 | 0 | 9
  Number of Severe TEAEs | 88 | 23 | 101
  Number of TEAEs with AZD1775 discontinued | 3 | 0 | 3
  Number of TEAEs with paclitaxel discontinued | 1 | NA — Patients in Cohort 1a did not receive paclitaxel. | 3
  Number of TEAEs with carboplatin discontinued | 0 | 0 | 3
  Number of TEAEs with fatal outcome | 1 | 0 | 2
  Number of Dose-Limiting Toxicities (DLT) | 1 | 1 | 2
  Number of TEAEs with DLT | 1 | 1 | 2

3. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events During AZD1775 Monotherapy Cycle by System Organ Class and Preferred Term
Description: The number of patients with TEAEs during AZD1775 Monotherapy Cycle was analyzed in the safety analysis set which was comprised of all patients who received at least one dose of the investigational drug.
Time Frame: Up to 1 week
Population: All patients who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 6 | 6
Participants
  Patients with at least 1 TEAE in AZD1775 cycle | 1 | 1 | 2
  Gastrointestinal Disorders - Nausea | 1 | 1 | 1
  Gastrointestinal Disorders - Constipation | 0 | 0 | 1
  Gastrointestinal Disorders - Diarrhoea | 0 | 1 | 0
  Immune System Disorders - Hypersensitivity | 0 | 0 | 1

4. Primary Outcome: Number of Patients With Clinically Important Changes in Haematology and Coagulation TEAEs by System Organ Class and Preferred Term
Description: The number of patients with clinically important changes in haematology and coagulation TEAEs was analyzed in the safety analysis set which was comprised of all patients who received at least one dose of the investigational drug.
Time Frame: Up to 21 days (1 Cycle)
Population: All patients who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 6 | 6
Participants
  Blood & Lymphatic System Disorders (BLSD) Anaemia | 6 | 4 | 5
  BLSD - Neutropenia | 3 | 0 | 2
  BLSD - Thrombocytopenia | 1 | 1 | 2
  BLSD - Febrile Neutropenia | 1 | 0 | 2
  Investigations - WBC Count Decreased | 5 | 3 | 5
  Investigations - Neutrophil Count Decreased | 3 | 4 | 3
  Investigations - Platelet Count Decreased | 4 | 3 | 3
  Investigations - Haematocrit Decreased | 1 | 0 | 0
  Investigations - Monocyte Count Decreased | 1 | 0 | 0

5. Primary Outcome: Number of Patients With Clinically Important Abnormalities in Clinical Chemistry by Preferred Term
Description: The number of patients with clinically important changes in clinical chemistry TEAEs was analyzed in the safety analysis set which was comprised of all patients who received at least one dose of the investigational drug.
Time Frame: Up to 21 days (1 Cycle)
Population: All patients who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 6 | 6
Participants
  Aspartate aminotransferase increased | 0 | 2 | 1
  Alanine aminotransferase increased | 0 | 1 | 0
  Blood alkaline phosphatase increased | 1 | 0 | 0
  Blood lactate dehydrogenase increased | 1 | 0 | 0
  C-reactive protein increased | 1 | 0 | 0
  Hypoalbuminemia | 2 | 0 | 2
  Hypokalemia | 1 | 1 | 2
  Hypophosphatemia | 1 | 0 | 2
  Dehydration | 1 | 0 | 1
  Hyperglycaemia | 2 | 0 | 0
  Hypocalcaemia | 0 | 0 | 1
  Hyponatraemia | 1 | 0 | 1
  Hypercalcaemia | 0 | 0 | 1
  Hypercholsterolaemia | 0 | 0 | 1
  Hypoglycaemia | 1 | 0 | 0
  Hypomagnesaemia | 0 | 0 | 1
  Azotemia | 1 | 0 | 0
  Hepatic function abnormal | 1 | 0 | 0

6. Primary Outcome: Number of Patients With Clinically Important Abnormalities in Vital Signs by Preferred Term
Description: The number of patients with clinically important changes in vital sign TEAEs was analyzed in the safety analysis set which was comprised of all patients who received at least one dose of the investigational drug.
Time Frame: Up to 21 days (1 Cycle)
Population: All patients who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 6 | 6
Participants
  Pyrexia | 3 | 1 | 4
  Hypotension | 2 | 0 | 1

7. Secondary Outcome: Best Overall Response
Description: The number of subjects with best overall response in CR, PR, NE, SD, PD subcategory. Best overall response is calculated based on the overall visit responses from each RECIST assessment.
Time Frame: Up to 18 months
Population: Best overall response was analyzed in the Evaluable-for-Response set, comprised of all patients who received at least one dose of the investigational drug and who had measurable disease at baseline.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Partial Response | 1 | 1 | 3
  Not Evaluable | 1 | 2 | 1
  Stable Disease | 2 | 2 | 2
  Progressive Disease | 2 | 1 | 0
  Complete Response | 0 | 0 | 0

8. Secondary Outcome: Number of Patients With an Objective Response
Description: Objective response is defined as either a complete response or a partial response.
Time Frame: Up to 18 months
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 1 | 3

9. Secondary Outcome: Percentage of Patients With an Objective Response
Description: Objective response is defined as either a complete response or a partial response.
Time Frame: Up to 18 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
Percentage | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 50 [11.8 to 88.2]

10. Secondary Outcome: Number of Patients With Clinical Benefit
Description: Clinical benefit is defined as achieving complete response, partial response, or stable disease.
Time Frame: Up to 18 months
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
Participants | 3 | 3 | 5

11. Secondary Outcome: Percentage of Patients With Clinical Benefit
Description: Clinical benefit is defined as achieving complete response, partial response, or stable disease.
Time Frame: Up to 18 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
Percentage | 50 [11.8 to 88.2] | 50 [11.8 to 88.2] | 83.3 [35.9 to 99.6]

12. Secondary Outcome: Duration of Response
Description: The duration of response is defined as the time in weeks from the date of first documented overall response occurrence of CR or PR, (whichever was recorded first) to the earliest date that progressive disease/death was documented. If progression or death has not been documented, a patient's DoR was censored at the date of last tumour assessment.
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
Weeks | 18.1 [0.00 to 9999.9] | 0.00 [0.00 to 9999.9] | 20.7 [0.00 to 9999.9]

13. Secondary Outcome: Peak Plasma Concentration (Cmax) of AZD1775 Following Single Dose Administration of AZD1775 Monotherapy
Time Frame: PK Samples collected in all treatment groups on Cycle 0 Day 1, Cycle 1 Day 1, and Cycle 1 Day 3 before the first (morning) dose of AZD1775 (predose) and at 1, 2, 4, 6, and 8 hours postdose
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 4 | 6
nM | 689.1 (51.79) | 649.2 (10.74) | 1066 (38)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of AZD1775 Following Single Dose Administration of AZD1775 Monotherapy
Time Frame: PK Samples will be collected in all treatment groups on Cycle 0 Day 1, Cycle 1 Day 1, and Cycle 1 Day 3 before the first (morning) dose of AZD1775 (predose) and at 1, 2, 4, 6, and 8 hours postdose
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 7 | 5 | 6
hours | 2.02 [1.00 to 8.00] | 3.95 [2.00 to 8.00] | 3.96 [1.00 to 5.87]

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Time of the Last Measurable Concentration (AUC0-t) Following Single Dose Administration of AZD1775 Monotherapy
Time Frame: as for outcome 14
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 4 | 6
nM*h | 3521 (44.91) | 3387 (12.54) | 5331 (37.42)

16. Secondary Outcome: Plasma Concentration of AZD1775 8 Hours After Single Dose Administration (C8h) of AZD1775 Monotherapy
Time Frame: as for outcome 14
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 4 | 6
nM | 370.1 (29.15) | 343.5 (29.97) | 612 (36.6)

17. Secondary Outcome: Peak Plasma Concentration (Cmax) of AZD1775 Following Oral Dose of AZD1775 in Combination With IV Infusion of Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: AZ1775:C0D1, C1D1, & C1D3 before AZD1775 dose and at 1,2,4,6&8 hrs postdose. Paclitaxel:C1D1 before paclitaxel infusion & at 1.5,3,4,6&8 hrs after start of infusion Carboplatin:C1D1 before carboplatin infusion &at 1,2,4,6&8 hrs after start of infusion
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 5 | 5 | 6
nM | 705.4 (28.03) | 654.8 (32.27) | 1133 (16.3)

18. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of AZD1775 Following Single Dose of AZD1775 in Combination With IV Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
hours | 4.00 [0.95 to 8.02] | 4.04 [3.98 to 6.00] | 4.00 [2.05 to 4.08]

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Time of the Last Measurable Concentration (AUC0-t) Following Single Dose of AZD1775 in Combination With IV Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 5 | 5 | 6
nM*h | 4191 (34.89) | 2902 (33.21) | 5606 (20.02)

20. Secondary Outcome: Plasma Concentration of AZD1775 8 Hours After Single Dose Administration (C8h) of AZD1775 in Combination With IV Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
nM | 444.6 (27.83) | 378.2 (27.61) | 805.9 (27.5)

21. Secondary Outcome: Peak Plasma Concentration (Cmax) of AZD1775 at Steady State When Given in Combination With IV Infusion of Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 5
nM | 1271 (30.52) | 1129 (25.51) | 2289 (32.82)

22. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of AZD1775 at Steady State When Given in Combination With IV Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
hours | 4.00 [2.05 to 4.08] | 3.09 [1.95 to 4.08] | 4.04 [1.00 to 7.95]

23. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Time of the Last Measurable Concentration (AUC0-t) at Steady State for AZD1775 in Combination With IV Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 5
nM*h | 8300 (32.85) | 7154 (32.29) | 14870 (34.05)

24. Secondary Outcome: Plasma Concentration of AZD1775 8 Hours After Administration (C8h) at Steady State in Combination With IV Paclitaxel and Carboplatin (Cohorts 1 and 2) or Carboplatin Alone (Cohort 1a)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 6 | 6
nM | 982 (30.17) | 774.6 (32.96) | 1700 (37.6)

25. Secondary Outcome: Peak Plasma Concentration (Cmax) of Paclitaxel Following Single IV Infusion in Combination With Single Dose Oral AZD1775 and IV Carboplatin
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 0 | 4
ng/mL | 4848 (31.13) |  | 5361 (4.744)

26. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC0-t) of Paclitaxel Following Single IV Infusion in Combination With Single Dose Oral AZD1775 and IV Carboplatin
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 0 | 4
h*ng/mL | 13100 (36.11) |  | 16360 (20.11)

27. Secondary Outcome: Plasma Concentration of Paclitaxel at the End of Infusion (Ceoi) When Given Combination With Oral AZD1775 and IV Carboplatin.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 0 | 4
ng/mL | 4791 (32.33) |  | 5361 (4.744)

28. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of IV Paclitaxel When Given in Combination With Oral AZD1775 and IV Carboplatin
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 0 | 4
hours | 2.99 [1.55 to 3.08] |  | 3.03 [3.02 to 3.10]

29. Secondary Outcome: Time to Last Detectable Concentration (Tlast) of Paclitaxel When Given in Combination With Oral AZD1775 and IV Carboplatin
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 0 | 4
hours | 2.99 [1.55 to 3.08] |  | 3.03 [3.02 to 3.10]

30. Secondary Outcome: Peak Plasma Concentration (Cmax) of Platinum Following Single IV Infusion of Carboplatin Over 1 Hour in Combination With Single Oral Dose AZD1775 Alone (Cohort 1a) or With IV Paclitaxel (Cohorts 1 and 2)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 4 | 3
ng/mL | 13300 (17.41) | 18550 (19.87) | 17500 (34.93)

31. Secondary Outcome: Area Under Plasma Concentration-time Curve From 0 to Last Measurable Conc. (AUC0-t) of Platinum Following Single IV Infusion of Carboplatin Over 1 Hour in Combination With Single Oral Dose AZD1775 Alone (Cohort 1a) or With IV Paclitaxel (Cohorts 1 & 2)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 4 | 3
h*ng/mL | 39370 (7.027) | 44630 (2.552) | 51340 (12.24)

32. Secondary Outcome: Plasma Concentration of Platinum at the End of Infusion (Ceoi) When Given as a 1 Hour Infusion in Combination With Oral AZD1775 and IV Paclitaxel.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 4 | 3
ng/mL | 13300 (17.41) | 18550 (19.87) | 17500 (34.93)

33. Secondary Outcome: Time to Peak Plasma Concentration of Platinum (Tmax) When Given as a 1 Hour Infusion in Combination With Oral AZD1775 and IV Paclitaxel.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 4 | 3
hours | 1.02 [1.02 to 1.10] | 1.02 [1.00 to 1.03] | 1.02 [1.00 to 1.02]

34. Secondary Outcome: Time to Last Detectable Concentration of Platinum (Tlast) When Given as a 1 Hour Infusion in Combination With Oral AZD1775 and IV Paclitaxel.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 4 | 3
hours | 7.98 [7.83 to 8.00] | 7.28 [7.20 to 7.98] | 8.00 [7.83 to 8.08]

35. Secondary Outcome: Peak Plasma Concentration (Cmax) of Platinum Following Single IV Infusion of Carboplatin Over 2 Hours in Combination With Single Oral Dose AZD1775 Alone (Cohort 1a) or With IV Paclitaxel (Cohorts 1 and 2)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 1 | 0
ng/mL | 15960 (26.51) | 13200 (0) |

36. Secondary Outcome: Area Under Plasma Concentration-time Curve From 0 to Last Measurable Conc. (AUC0-t) of Platinum Following Single IV Infusion of Carboplatin Over 2 Hours in Combination With Single Oral Dose AZD1775 Alone (Cohort 1a) or With IV Paclitaxel (Cohorts 1 & 2)
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 6 | 1 | 0
h*ng/mL | 56240 (17.2) | 48700 (0) |

37. Secondary Outcome: Plasma Concentration of Platinum at the End of Infusion (Ceoi) When Given as a 2 Hour Infusion in Combination With Oral AZD1775 and IV Paclitaxel.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 1 | 0
ng/mL | 15960 (26.51) | 12200 (0) |

38. Secondary Outcome: Time to Peak Plasma Concentration of Platinum (Tmax) When Given as a 2 Hour Infusion in Combination With Oral AZD1775 and IV Paclitaxel.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 1 | 0
hours | 1.97 [1.92 to 2.00] | 1.08 [1.08 to 1.08] |

39. Secondary Outcome: Time to Last Detectable Concentration of Platinum (Tlast) When Given as a 2 Hour Infusion in Combination With Oral AZD1775 and IV Paclitaxel.
Time Frame: as for outcome 17
Population: The pharmacokinetic analysis set consisted of all dosed patients for whom an adequate PK profile was obtained.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
Number analyzed (Participants) | 3 | 1 | 0
hours | 7.95 [7.92 to 8.03] | 8.00 [8.00 to 8.00] |

ADVERSE EVENTS:
Time Frame: Up to 18 months.
Arm/Group | Cohort 1 | Cohort 1a | Cohort 2
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/7 | 0/6 | 4/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 1a (N=6) | Cohort 2 (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 1a (N=6) | Cohort 2 (N=6)
Anaemia (Blood and lymphatic system disorders) | 6 (48) | 4 (21) | 5 (37)
Neutropenia (Blood and lymphatic system disorders) | 3 (18) | 0 (0) | 2 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (9) | 1 (6) | 2 (23)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Eyelid Oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (36) | 6 (27) | 5 (37)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (25) | 3 (13) | 4 (49)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 2 (4) | 2 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (20) | 4 (15) | 5 (27)
Oesphageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctologia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (7)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fatugue (General disorders) | 2 (3) | 2 (5) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (11) | 2 (4) | 4 (9)
Asthenia (General disorders) | 1 (2) | 1 (1) | 2 (4)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (7) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fallopian tube abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rash (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hematocrit decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (50) | 3 (29) | 3 (21)
White blood cell count decreased (Investigations) | 5 (26) | 3 (10) | 5 (31)
Blood alklaine phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (10) | 4 (8) | 3 (15)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (6) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 4 (10) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (12) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 2 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (6)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 2 (2) | 1 (2)
Peripheral neuropathy (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2) | 2 (5)
Azotemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (3)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ingrown nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (3)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In the secondary outcome measure Duration of Response for which data are reported as weeks (95% CI) several instances occurred where the 95% CI could not be calculated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No